CLINICAL TRIAL: NCT01346956
Title: Acute Cardiovascular Effects of Cigarette Smoking
Status: Completed | Type: Observational
Sponsor: Andhra Medical College (Other Government)
Responsible Party: Ravi Venkatachelam Chitrapu, Andhra Medical College
Other Study IDs: 02AMCRAVSAND07
Record Dates: First submitted 2011-05-02; First posted 2011-05-04 (Estimated); Last update posted 2011-05-04 (Estimated); Status verified 2003-01

CONDITIONS: Smoking
Keywords: Cigarette; Smoking; Cardiovascular Effects; 2D Echocardiography; Doppler
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Twenty healthy smokers will be subjected to measurement of Pulse, Blood Pressure, electrocardiogram (ECG) and Echo at baseline and after smoking a cigarette. The measurements will be compare for any cardiovascular effects of a cigarette smoking on these parameters.

DETAILED DESCRIPTION:
Twenty male persons habituated to smoking (at least 5 cigarettes/day) will be recruited after an informed consent. Healthy persons with no systemic illness will be included. After a history and a routine examination, subjects will be asked to abstain from smoking for 3 hours and then their pulse, BP, ECG and echo recorded. The measurements will be repeated after 15 min. and the average of these two taken as baseline readings. Then, they will be asked to smoke a cigarette and the measurements taken again. Special focus will be on Doppler measures of left ventricular (LV) function. The measurements are repeated immediately and at 5,10 and 15 min. The data will be analyzed for any cardiovascular effects of smoking a cigarette. Chi square test for proportions and t-test for means will be done. A p value < 0.05 will be taken as significant.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male smokers (at least 5 cigarettes /day) >18 years old.

Exclusion Criteria:

* Any cardiac or respiratory or systemic illness,including hypertension.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Twenty healthy male smokers
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2002-07; Primary Completion 2002-08 (Actual); Study Completion 2002-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Venkatachelam R Chitrapu, MD DM, Principal Investigator — Andhra Medical College
Locations (1):
- Andhra Medical College, Visakhapatnam, Andhra Pradesh, India